CLINICAL TRIAL: NCT05384730
Title: A Feasibility and Acceptability Study of a Virtual Multimodal Intervention Delivered by Volunteers to Improve Functional Outcomes of Frail Older Adults Discharged From Hospital
Brief Title: Frail2Fit Study: Online Nutrition and Exercise Support for Older Adults With Frailty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: Bournemouth University (Other); University of Southampton (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RHM MED1860 - Frail2Fit
Record Dates: First submitted 2022-05-17; First posted 2022-05-20 (Actual); Results first posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2024-10

CONDITIONS: Frailty; Malnutrition; Sedentary Behavior
MeSH Terms: conditions — Frailty; Malnutrition; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): This group will receive the weekly group exercise and nutrition support which will be delivered online by trained volunteers. The duration of the intervention is 12 weeks.
  Interventions: Other: Group nutrition and exercise support

INTERVENTIONS:
Other: Group nutrition and exercise support — Weekly group nutrition and exercise support delivered online through trained volunteers

SUMMARY:
Frail2Fit will explore the feasibility of training volunteers to deliver online nutrition, exercise, and behaviour change (supported self-management) to improve the health of older people after discharge from hospital. The study also aims to explore if the supported self-management is acceptable to older people, their family members and/or carers, and the volunteers.

Between 30-60% of older people in hospital lose muscle strength and function (deconditioning) and around 14% of older adults in hospital are frail. Reduced muscle function and frailty increase risk of poor health outcomes, including reduced quality of life, increased risk of hospital readmission and increased risk of mortality. Therefore, intervening to prevent functional decline is a high-priority patient-centred outcome. Current evidence suggest that physical activity (PA) and nutrition interventions are key to maintaining independence and improving frailty status. In response to the COVID-19 restrictions, healthcare and rehabilitation have increasingly turned to virtual modes of delivery, such as telehealth methods. The increasing use of technology in the daily lives of many allows PA and nutrition interventions to be delivered online. For instance, the investigators have developed and evaluated a programme using online clinics to successfully support over 600 cancer patients living at home to stay active and eat well with provision of emotional support (SafeFit study). With many older people now using the internet for social connection, the team have an opportunity to investigate whether a similar model can improve the health of older people.

This study aims to explore the feasibility and acceptability of implementing volunteer-led online exercise and nutrition support to frail older people discharged from hospital. The investigators aim to develop and evaluate a training programme for volunteers, determine the acceptability of the intervention through qualitative methods and identify facilitators and barriers to its implementation. The investigators will also explore the impact of the intervention on health outcomes for older people to inform future trial.

DETAILED DESCRIPTION:
Study design A quasi-experimental mixed methods approach will be used to determine the feasibility and acceptability of implementing a volunteer-led multi-modal intervention for discharged older adults with frailty. This feasibility study will be conducted at the University Hospital Southampton NHS Foundation Trust (UHS), training hospital volunteers to deliver virtual group support for older adults discharged from UHS. The acceptability of the intervention will also be examined through qualitative interviews to explore the views and experiences of volunteers, trainers, carers and older adults involved in this study. The impact of the intervention on physical activity levels and functional outcomes will be measured.

Participants Older adults aged 65 years or above with frailty (clinical frailty score ≥5) who have been discharged from UHS will be invited to participate in this study. Participants must be able to walk at least a few steps upon hospital discharge and be cleared by their clinician as safe to exercise. Patients will be identified and approached by their clinical care team, if they are interested in participating in the research a member of the research team will obtain written informed consent. A sample size of 30 participants was chosen in line with previous sample size recommendations for feasibility studies of 24-50 participants. This sample size was considered an appropriate number that is pragmatic and achievable within the study timescale and resources available.

Recruitment and training of volunteers Volunteers from the UHS patient support hub will be invited to participate in the study and receive training to deliver the intervention. Volunteers aged 16 years or above who have completed the generic volunteer clearance and training at the hospital and who are safe to exercise will be identified by hospital voluntary services. Interested volunteers will be approached by a member of the research team to complete written informed consent. A sample size of 6 volunteers was chosen to provide sufficient cover to deliver the Frail2Fit intervention to small groups of older adults with 2 volunteers supporting each group.

The volunteer training programme will consist of a bespoke training package adapted from the SafeFit training guidance, supported, and delivered by an expert dietician (Prof Jane Murphy), psychologist (Judit Varkonyi-Sepp), and clinical exercise instructor, Dr Samantha Meredith (SM), and led by the PI, Dr Stephen Lim (SL). Training will be conducted at UHS for 2 days and 1 day of online training. The training sessions will include training on personal safety and safety of participants, and the exercise, nutrition and behaviour change protocols. As these are existing volunteers, they would have been recruited, and received the generic clearance and training provided by UHS. Throughout the study period, fidelity checks will be conducted by SM and SL to ensure that the volunteers are delivering high quality exercise sessions. Volunteers will also receive training on how to document adverse events that occur during the classes.

Intervention The intervention duration will be 3 months. Participants will receive three group sessions per week for 1 month (weeks 1-4), twice per week for the second month (weeks 5-8), and once weekly for the last month (weeks 9-12), with a maximum of 24 sessions. The tapered nature of the intervention was chosen to provide suitable support for older adults post-discharge with the aim to gradually encourage increased self-management to foster independence post-intervention. Components of the intervention, including exercise, nutrition support and behaviour change support, will be delivered from an online platform (Zoom). Each group session will last 40-60 minutes, including 20-30 minutes of exercise followed by 20-30 minutes of nutrition support. The components of the intervention and the training package have been adapted from the SafeFit trial and will be delivered in line with behaviour change principles to maximise participant uptake, adherence and lifestyle self-management.

The exercise will consist of volunteer-led group progressive resistance exercise training for 20-30 minutes. To align with home-based safety considerations, the exercises will be performed seated. Seated exercise will focus on strengthening upper and lower limbs (8 major muscle groups) and enhancing whole body range of motion and flexibility, tailored specifically to meet the needs of older adults and to minimise the risks of injury.

The nutrition component will involve reviewing patient diet and eating habits using the Nutrition Wheel to ensure nutrition is appropriate and patients are not at risk of undernutrition. The Nutrition Wheel is an interactive tool developed from the Patients Association Nutrition Checklist and used to engage individuals in conversation about unintentional weight loss and malnutrition.

Healthy conversation skills (HCS) guided by principles of Making Every Contact Count (MECC) will be used to support the delivery of the exercise and nutrition components in the current intervention. The MECC approach supports positive behaviour change through encouraging client-centred brief conversations surrounding health and well-being. Training will enable volunteers to have the confidence and competence to deliver healthy lifestyle messages to empower participants.

Data collection Participant characteristics including age, gender, domicile status, weight, body mass index, malnutrition status (MUST), baseline nutritional status (e.g., use of nutritional supplements and dietician support), co-morbidities (Charlson Co-morbidity Index), cognition (Mini-mental state examination; MMSE) and number of medications will be recorded. Volunteer characteristics recorded will include age, occupation, qualifications, volunteering experience, and employment status.

The primary outcome measures are feasibility and acceptability of the intervention. The feasibility of implementing a volunteer-led online multi-modal intervention will be assessed by determining the number of volunteers recruited, trained and retained at the end of the study, the number of intervention sessions delivered and fidelity of volunteer delivery. Moreover, participant recruitment, retention and adherence to the intervention will be measured, as well as any adverse events. Interviews will be conducted among older adults (N= 6), volunteers (N= 6), and those involved in recruiting participants and training volunteers (N= 3), to determine the acceptability of the intervention and to explore barriers and enablers to the implementation of the intervention. Interviews will be semi-structured to help guide conversation whilst allowing participants the flexibility to elaborate and reflect on any meaningful experiences.

The secondary outcomes will include the measurement of physical activity levels (PASE and GENE Activ accelerometer), physical function (Bathel), appetite (SNAQ), well-being (WEMWBS), anxiety and depression (HADS), quality of life (EQ-5D-5L ), and self-efficacy for managing chronic disease. These will be measured at baseline (in hospital), 3 months (via telephone) and 6 months (via telephone).

Data analysis Quantitative data analysis Data collected will be double entered into a secured database for analysis. Statistical analysis will be conducted using the statistical software SPSS. Descriptive statistics -median (IQR); mean (SD); number (%) - will be used to analyse the numbers of volunteers recruited, trained and retained, as well as the type and extent of progression of the resistance exercise, and duration of their activity, and patients' adherence to the intervention. Analysis of the above outcome measures will be used to develop an assessment of the feasibility of delivering this intervention. To determine suitability for a future, fully-powered effectiveness study of the intervention, outcome measures recorded at baseline will be compared to measurement at 3 and 6 months to determine if the intervention had an impact on physical activity levels measured by PASE and GENEActiv, functional outcomes including Barthel, SNAQ, HADS, WENWBS, self-efficacy and EQ-5D-5L. The distribution of each outcome measure will be assessed for normality and described using parametric or non-parametric statistics accordingly. A basic cost-analysis of the training programme will be carried out, costing the time of clinical staff involved in delivering the training.

Qualitative data analysis Data collected from the interviews will be transcribed verbatim and analysed using thematic analysis (TA). The audio-recordings will be transcribed by an administrative colleague within the research department who is experienced in transcribing qualitative data. TA is a method for identifying, analysing and reporting patterns or themes within data and is widely used in qualitative research. There are six phases in the process of conducting TA: Phase 1 - familiarising with the data, Phase 2 - generating initial codes, Phase 3 - searching for themes, Phase 4 - reviewing themes, Phase 5 - defining and naming themes, and Phase 6 - producing the report. Analysis of qualitative data will be conducted using either Microsoft Word, or with the help of NVIVO, depending on the amount of data collected. Transcribed text will be read and coded separately and then together by two researchers. The codes will be analysed to generate concepts and ideas to determine the acceptability of the intervention, and to identify facilitators and barriers to the implementation process. The codes act as tags or labels to help catalogue key concepts embedded within the raw data. From the codes, themes will be developed to reflect the views and experiences of the community-dwelling older adults and volunteers regarding the community-based PA intervention.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Older adults age 65 years and above
* Able to provide written consent
* Discharged from UHS
* Identified as frail (Clinical Frailty Scale ≥5)
* Able to walk at least a few steps upon hospital discharge
* Able to communicate fluently enough in English

Volunteers:

* Established volunteers at UHS patient support hub
* Age 16 years and above
* Completed the generic volunteer clearance and training at UHS
* Able to provide written informed consent
* Able to communicate fluently enough in English

Exclusion Criteria:

Patients:

* Older adults who are not able to safely complete the exercises included in the intervention
* Patients who are discharged to rehabilitation units, or care homes
* Patients receiving end of life care

Volunteers:

- Volunteers who are unable to safely complete the exercises included in the intervention will be excluded from the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-10-28 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2024-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen ER Lim, PhD, Principal Investigator — University of Southampton
Locations (1):
- University Hospital Southampton, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grimmett C, Bates A, West M, Leggett S, Varkonyi-Sepp J, Campbell A, Davis J, Wootton S, Shaw C, Barlow R, Ashcroft J, Scott A, Moyes H, Hawkins L, Levett DZH, Williams F, Grocott MPW, Jack S. SafeFit Trial: virtual clinics to deliver a multimodal intervention to improve psychological and physical well-being in people with cancer. Protocol of a COVID-19 targeted non-randomised phase III trial. BMJ Open. 2021 Aug 26;11(8):e048175. doi: 10.1136/bmjopen-2020-048175. PMID 34446487
- [Background] Lim SER, Meredith S, Agnew S, Clift E, Ibrahim K, Roberts H. Evaluating the feasibility and acceptability of virtual group exercise for older adults delivered by trained volunteers: the ImPACt study protocol. BMJ Open. 2022 Feb 1;12(2):e052631. doi: 10.1136/bmjopen-2021-052631. PMID 35105576
- [Background] Meredith SJ, Roberts H, Grocott MPW, Jack S, Murphy J, Varkonyi-Sepp J, Bates A, Lim SER. Frail2Fit study protocol: a feasibility and acceptability study of a virtual multimodal intervention delivered by volunteers to improve functional outcomes in older adults with frailty after discharge from hospital. BMJ Open. 2023 Mar 16;13(3):e069533. doi: 10.1136/bmjopen-2022-069533. PMID 36927597

RESULTS

PARTICIPANT FLOW:
Groups:
- Hospital Volunteers: Hospital volunteers trained to deliver the Frail2Fit intervention
Period: Overall Study
Arm/Group | Intervention Arm | Hospital Volunteers
Started | 27 | 5
Completed | 17 | 3
Not Completed | 10 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Lack of social support | 2 | 0
Not completed — Hospital readmission | 2 | 0
Not completed — Disease progression | 5 | 0
Not completed — Overwhelmed with College commitments | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Hospital Volunteers: Hospital volunteers were trained to deliver the Frial2Fit intervention
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Hospital Volunteers | Total
Number analyzed (Participants) | 27 | 5 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Baseline characteristics were not collected for 1 participant who underwent an operation and moved wards
  years
    number analyzed (Participants) | 26 | 5 | 31
    (all) | 80.3 (7) | 16.4 (0.49) | 70 (24.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 3 | 18
  Male | 12 | 2 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: One enrolled participant withdrew from the study before their baseline data collections were completed
  Participants
    Ethnicity: number analyzed (Participants) | 26 | 5 | 31
    Ethnicity: White British | 26 | 2 | 28
    Ethnicity: Polish | 0 | 1 | 1
    Ethnicity: Asian British | 0 | 1 | 1
    Ethnicity: Chinese | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 27 | 5 | 32
Cognitive status (Mini Mental State Examination) [Median (Inter-Quartile Range); unit: units on a scale] — The mini mental state examination assesses cognitive status with scores ranging from 0-30. A higher score indicates better cognitive status than a lower score. A score of 0-17 indicates severe cognitive impairment, 18-23 indicates mild cognitive impairment, and 24-30 indicates no cognitive impairment. Population: Baseline characteristics in the intervention group were not collected for 1 participant who underwent an operation and moved wards. We were only interested in measuring this characteristic for the intervention group and not the volunteers.
  units on a scale
    number analyzed (Participants) | 26 | 0 | 26
    (all) | 28 [24.8 to 29] |  | 28 [24.8 to 29]
Charlson comorbidity index [Median (Inter-Quartile Range); unit: units on a scale] — The Charlson Comorbidity Index (CCI) predicts the mortality for a patient who may have a range of concurrent conditions (comorbidities), such as heart disease, AIDS, or cancer (considering a total of 17 categories). Scores range from 1-9, with a higher score indicating greater risk of mortality. Population: Baseline characteristics were not collected for 1 participant who underwent an operation and moved wards. We were only interested in measuring this characteristic for the intervention group and not the volunteers.
  units on a scale
    number analyzed (Participants) | 26 | 0 | 26
    (all) | 4 [4 to 5.3] |  | 4 [4 to 5.3]
Clinical frailty scale [Median (Inter-Quartile Range); unit: units on a scale] — The clinical frailty scale is a tool to screen for and assess frailty, ranging from 1 very fit through to 9 terminally ill. Frailty is considered when a person has a score of 5 or more.
  1. very fit
  2. well
  3. managing well
  4. vulnerable
  5. mildly frail
  6. moderately frail
  7. severly frail
  8. very severly frail
  9. terminally ill Population: Baseline characteristics were not collected for 1 participant who underwent an operation and moved wards. We were only interested in measuring this characteristic for the intervention group and not the volunteers.
  units on a scale
    number analyzed (Participants) | 26 | 0 | 26
    (all) | 6 [5 to 6] |  | 6 [5 to 6]
Number of medications [Median (Inter-Quartile Range); unit: count] — Population: Baseline characteristics were not collected for 1 participant who underwent an operation and moved wards. We were only interested in measuring this characteristic for the intervention group and not the volunteers.
  count
    number analyzed (Participants) | 26 | 0 | 26
    (all) | 9 [6 to 11.3] |  | 9 [6 to 11.3]
Length of hospital stay [Median (Inter-Quartile Range); unit: days] — Population: Baseline characteristics were not collected for 1 participant who underwent an operation and moved wards. We were only interested in measuring this characteristic for the intervention group and not the volunteers.
  days
    number analyzed (Participants) | 26 | 0 | 26
    (all) | 15 [8.8 to 22.5] |  | 15 [8.8 to 22.5]
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] — Body mass index is calculated by dividing an adult's weight in kilograms by their height in metres squared.
  under 18.5 - This is described as underweight. between 18.5 and 24.9 - This is described as the 'healthy range'. between 25 and 29.9 - This is described as overweight between 30 and 39.9 - This is described as obesity 40 or over - This is described as severe obesity Population: Baseline characteristics were not collected for 1 participant who underwent an operation and moved wards. We were only interested in measuring this characteristic for the intervention group and not the volunteers.
  kg/m^2
    number analyzed (Participants) | 26 | 0 | 26
    (all) | 25.5 [20.7 to 28] |  | 25.5 [20.7 to 28]

OUTCOME MEASURES:

1. Primary Outcome: Volunteers Trained
Description: The number of volunteers recruited to the study and trained.
Time Frame: 6 months
Population: Does not apply to intervention group
Measure: Count of Participants; unit: Participants
Groups:
- Hospital Volunteers: Hospital volunteers were trained to deliver the frail2fit intervention
Arm/Group | Intervention Arm | Hospital Volunteers
Number analyzed (Participants) | 0 | 5
Participants |  | 5

2. Primary Outcome: Volunteer Retention
Description: The number of volunteers retained at the end of the study
Time Frame: 6 months
Population: This measure was not applicable for the intervention group
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Hospital Volunteers
Number analyzed (Participants) | 0 | 5
Participants |  | 3

3. Primary Outcome: Adherence - Online
Description: The percentage of online sessions completed
Time Frame: post-intervention = 3-months
Population: This measure is not applicable for the hospital volunteer group
Measure: Median (Inter-Quartile Range); unit: percentage of completed sessions
Arm/Group | Intervention Arm | Hospital Volunteers
Number analyzed (Participants) | 17 | 0
percentage of completed sessions | 75 [38 to 92] |

4. Primary Outcome: Adherence - Telephone Support
Description: The percentage of telephone sessions completed
Time Frame: post-intervention= 3-months
Population: This measure is not applicable for the hospital volunteer group
Measure: Median (Inter-Quartile Range); unit: percentage of completed sessions
Arm/Group | Intervention Arm | Hospital Volunteers
Number analyzed (Participants) | 17 | 0
percentage of completed sessions | 80 [68.5 to 94.5] |

5. Secondary Outcome: Device-based Physical Activity Levels
Description: Device-based physical activity was measured using wrist-worn GENEActiv accelerometers, including light-physical activity, moderate-vigorous physical activity, and sedentary time (mins/day).
Time Frame: Baseline, post-intervention (3-months) and follow-up (6-months)
Population: This measure is not applicable for the hospital volunteer group
Measure: Mean (Standard Deviation); unit: mins/day
Groups:
- Baseline - Intervention Arm: This group will receive the weekly group exercise and nutrition support which will be delivered online by trained volunteers. The duration of the intervention is 12 weeks.
  Group nutrition and exercise support: Weekly group nutrition and exercise support delivered online through trained volunteers - Repeated measures design - baseline
- Post-Intervention (3-month): Frail2Fit intervention group - repeated measures design - timeframe: post-intervention
- Follow-Up (6-month): Frail2Fit intervention repeated measures - 3-month follow-up of data
Arm/Group | Baseline - Intervention Arm | Post-Intervention (3-month) | Follow-Up (6-month) | Hospital Volunteers
Number analyzed (Participants) | 17 | 17 | 17 | 0
mins/day
  Light physical activity | 29.95 (21.07) | 38.88 (24.98) | 33.37 (24.67) |
  Moderate-vigorous physical activity | 18.72 (17.25) | 23.08 (18.87) | 21.02 (18.12) |
  Inactive/sedentary time | 751.42 (51.86) | 744.39 (43.84) | 731.01 (52.69) |
Statistical Analysis 1: Comparison: Baseline - Intervention Arm vs Post-Intervention (3-month) vs Follow-Up (6-month); Light physical activity compared overtime; Test type: Superiority; p = 0.10, ANOVA
Statistical Analysis 2: Comparison: Baseline - Intervention Arm vs Post-Intervention (3-month) vs Follow-Up (6-month); Moderate-vigorous physical activity compared overtime; Test type: Superiority; p = 0.30, ANOVA
Statistical Analysis 3: Comparison: Baseline - Intervention Arm vs Post-Intervention (3-month) vs Follow-Up (6-month); Inactive/sedentary time compared overtime; Test type: Superiority; p = 0.18, ANOVA

6. Secondary Outcome: Functional Ability
Description: The Barthel Index scores 10 items describing activities of daily living and mobility, with a higher number being a reflection of greater ability to function independently following hospital discharge. Scores range from 0-20.
Time Frame: Baseline, post-intervention (3-months) and follow-up (6-months)
Population: This measure is not applicable for the hospital volunteer group
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Baseline - Intervention Arm | Post-Intervention (3-month) | Follow-Up (6-month) | Hospital Volunteers
Number analyzed (Participants) | 17 | 17 | 17 | 0
units on a scale | 18 [14 to 20] | 19 [17.5 to 20] | 20 [16.5 to 20] |
Statistical Analysis 1: Comparison: Baseline - Intervention Arm vs Post-Intervention (3-month) vs Follow-Up (6-month); Test type: Superiority; p = 0.14, Chi-squared

7. Secondary Outcome: Appetite
Description: Simplified Nutritional Appetite Questionnaire (SNAQ). SNAQ is a four-item tool assessing appetite, satiety, taste of food and number of meals per day. SNAQ has a minimum score of 4 and a maximum score of 20, with a score of ≤14 indicating poor appetite.
Time Frame: Baseline, Post-intervention (3-month) and follow-up (6-month)
Population: This measure is not applicable for the hospital volunteer group
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline - Intervention Arm | Post-Intervention (3-month) | Follow-Up (6-month) | Hospital Volunteers
Number analyzed (Participants) | 17 | 17 | 17 | 0
score on a scale | 14.2 (3.3) | 15.4 (2.3) | 15.6 (2) |
Statistical Analysis 1: Comparison: Baseline - Intervention Arm vs Post-Intervention (3-month) vs Follow-Up (6-month); Test type: Superiority; p = 0.01, ANOVA

8. Secondary Outcome: Well-being
Description: Warwick-Edinburgh Well-Being Scale (WEMWBS). WEMWBS comprises 14 positively worded items relating to different aspects of positive mental health, including positive affect, satisfying interpersonal relationships and positive functioning. Each item is scored on a 5-point Likert scale from 1 (none of the time) to 5 (all of the time), with a higher score indicating a higher level of mental well-being. Total calculated scores range from 14-70.
Time Frame: Baseline, Post-intervention (3-month) and follow-up (6-month)
Population: This measure is not applicable for the hospital volunteer group
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline - Intervention Arm | Post-Intervention (3-month) | Follow-Up (6-month) | Hospital Volunteers
Number analyzed (Participants) | 17 | 17 | 17 | 0
score on a scale | 49.5 (8.2) | 50.2 (9.3) | 51.4 (9.6) |
Statistical Analysis 1: Comparison: Baseline - Intervention Arm vs Post-Intervention (3-month) vs Follow-Up (6-month); Test type: Superiority; p = 0.50, ANOVA

9. Secondary Outcome: Depression and Anxiety
Description: The Hospital Anxiety and Depression Scale (HADS). HADS comprises seven questions for anxiety and seven questions for depression. A score of 0-7 is normal, 8-10 borderline abnormal, and 11-21 abnormal. Scores can range from a minimum of 0 to a maximum of 21.
Time Frame: Baseline, post-intervention (3-month) and follow-up (6-month)
Population: This measure is not applicable for the hospital volunteer group
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Baseline - Intervention Arm | Post-Intervention (3-month) | Follow-Up (6-month) | Hospital Volunteers
Number analyzed (Participants) | 17 | 17 | 17 | 0
score on a scale
  Depression | 6 [3.5 to 8] | 3 [1 to 5] | 4 [3 to 7] |
  Anxiety | 4 [2 to 6.5] | 4 [2 to 6.5] | 4 [2.5 to 6] |
Statistical Analysis 1: Comparison: Baseline - Intervention Arm vs Post-Intervention (3-month) vs Follow-Up (6-month); Comparing depression scores overtime; Test type: Superiority; p = 0.03, Chi-squared
Statistical Analysis 2: Comparison: Baseline - Intervention Arm vs Post-Intervention (3-month) vs Follow-Up (6-month); Comparing anxiety scores overtime; Test type: Superiority; p = 0.96, Chi-squared

10. Secondary Outcome: Patient's Subjective Assessment of Quality of Life
Description: Quality of life was measured using the EuroQol (EQ-5D-5L) assessment comprising a short descriptive questionnaire. The questionnaire includes 5 domains (e.g., mobility; self-care; usual activities; pain/discomfort; and anxiety/depression) measured with 5 response levels from 'no problems' to 'extreme problems/unable'. A health state index score was calculated from individual health profiles using UK value set data (0.000 [minimum quality of life] - 1.000 [maximum quality of life]).
Time Frame: Baseline, Post-intervention (3-month) and follow-up (6-month)
Population: This measure is not applicable for the hospital volunteer group
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | Baseline - Intervention Arm | Post-Intervention (3-month) | Follow-Up (6-month) | Hospital Volunteers
Number analyzed (Participants) | 17 | 17 | 17 | 0
Score on a scale | 0.683 [0.489 to 0.708] | 0.733 [0.570 to 0.803] | 0.720 [0.456 to 0.813] |
Statistical Analysis 1: Comparison: Baseline - Intervention Arm vs Post-Intervention (3-month) vs Follow-Up (6-month); Test type: Superiority; p = 0.04, Chi-squared

11. Secondary Outcome: Self-efficacy for Managing Chronic Disease
Description: A 6-item scale will be used to assess participant's self-efficacy in managing their chronic disease. The scale contains items developed from the chronic disease self-management study covering domains, such as symptom control, role function, emotional functioning and communicating with health professionals. Each item is scored on a 10-point Likert scale from 1 (not at all confident) to 10 (totally confident). Higher scores indicate higher self-efficacy with scores ranging from 6-60.
Time Frame: Baseline, Post-intervention (3-month) and follow-up (6-month)
Population: This measure is not applicable for the hospital volunteer group
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Baseline - Intervention Arm | Post-Intervention (3-month) | Follow-Up (6-month) | Hospital Volunteers
Number analyzed (Participants) | 17 | 17 | 17 | 0
score on a scale | 37.4 (9.2) | 41.8 (6.5) | 40.9 (10.2) |
Statistical Analysis 1: Comparison: Baseline - Intervention Arm vs Post-Intervention (3-month) vs Follow-Up (6-month); Test type: Superiority; p = 0.13, ANOVA

12. Secondary Outcome: Self-reported Physical Activity
Description: Self-reported physical activity was measured using the physical activity scale for the elderly (PASE), which measures a broad spectrum of activities including leisure-time, household, and occupational PA during the previous 7 days. The PASE outcome is total self-reported physical activity which is scored from 0-400 with higher scores representing higher levels of physical activity.
Time Frame: Baseline, Post-Intervention (3-month), Follow-Up (6-months)
Population: This measure is not applicable for the hospital volunteer group
Measure: Mean (Standard Deviation); unit: PASE score on a scale
Arm/Group | Baseline - Intervention Arm | Post-Intervention (3-month) | Follow-Up (6-month) | Hospital Volunteers
Number analyzed (Participants) | 17 | 17 | 17 | 0
PASE score on a scale | 32.8 (35.2) | 50.8 (31.1) | 46.2 (39.8) |
Statistical Analysis 1: Comparison: Baseline - Intervention Arm vs Post-Intervention (3-month) vs Follow-Up (6-month); PASE analysis over time; Test type: Superiority; p = 0.01, ANOVA

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Intervention Arm | Hospital Volunteers
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/5
Other Adverse Events (participants affected / at risk) | 1/23 | 0/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Arm (N=23) | Hospital Volunteers (N=5)
Strained shoulder muscle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 — Participant receiving telephone support strained their shoulder muscle while using the resistance band during exercise training on the Frail2Fit intervention

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-03-13): https://cdn.clinicaltrials.gov/large-docs/30/NCT05384730/Prot_SAP_ICF_000.pdf